CLINICAL TRIAL: NCT01485978
Title: Early Prospective Therapy Trial to Delay Renal Failure in Children With Alport Syndrome
Brief Title: Efficacy and Safety Study to Delay Renal Failure in Children With Alport Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University Medical Center Goettingen (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EARLY_PRO-TECT_ALPORT
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Alport Syndrome; chronic kidney disease; renal fibrosis; nephroprotection; pediatric study
MeSH Terms: conditions — Renal Insufficiency, Chronic; Nephritis, Hereditary | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ramipril blinded (Active Comparator): oral treatment with 1 to 6 mg per body surface area ramipril once daily for 3 years
  Interventions: Drug: Ramipril
- placebo to ramipril (Placebo Comparator): Oral placebo treatment to ramipril once daily for 3 years or until progress to next disease level. After progression to next disease level, patients will be unblinded, and ramipril treatment will be initiated.
  Interventions: Drug: placebo to ramipril
- open label ramipril (Other): Open label treatment with ramipril as per protocol, if randomization is refused.
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — Ramipril (Delix) tablets containing 2.5 mg ramipril, oral application with 1 to 6 mg per body surface area ramipril once daily for 3 years.
  Arms: Ramipril blinded
Drug: placebo to ramipril — Oral application of placebo to ramipril, once daily with 1 to 6 mg per body surface area for 3 years or until disease progression.
  Arms: placebo to ramipril
Drug: Ramipril — Oral treatment with 1 to 6 mg per body surface area ramipril once daily for 3 years as per protocol.
  Arms: open label ramipril

SUMMARY:
This is a phase III, multi-centre, randomised, placebo-controlled, patient and investigator-blind study in paediatric patients with early stages of Alport syndrome to assess the safety and efficacy of the ACEi ramipril in slowing disease progression.

Alport syndrome stages that describe the extent of renal damage and loss of function are defined as:

* 0 Microhaematuria without microalbuminuria (usually at birth)
* I Microalbuminuria (30-300 mg albumin/gCrea)
* II Proteinuria >300 mg albumin/gCrea
* III > 25% decline of normal renal function (creatinine clearance)
* IV End stage renal failure (ESRF)

Eligible patients with Alport stages 0 and I will be randomly assigned at a 2:1 ratio to receive once daily ramipril or placebo. In addition, Alport stage II patients may be treated open Label. Eligible patients who, or whose parents/legal guardian refuse randomisation after eligibility is confirmed, and patients who have been treated with ramipril prior to the study, may be treated open-label with ramipril as per protocol. The total number of patients will not exceed 120, with the number of randomised patients not exceeding 60, and the number of patients treated open label from Day 1 of the study aimed to be approximately 60.

Randomised patients whose disease progresses to the next disease level during the 3 year treatment period will be unblinded, and open label ramipril treatment will be initiated and continued, respectively, depending on prior treatment randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Alport syndrome: Kidney biopsy (patient or affected relative/s), and/or mutation analysis (hemizygous X-chromosomal or homozygous autosomal-recessive) and assessment of criteria for clinical diagnosis (haematuria, positive family history regarding kidney diseases, ocular changes, labyrinthine hearing loss)
* Alport syndrome levels 0, I or II at screening (microhaematuria without microalbuminuria or microalbuminuria [30-300 mg albumin/gCrea]) or proteinuria >300 mg albumin/gCrea with GFR>80ml/min). Patients with Alport stage II are not subject to randomization but are treated opel label.
* Aged between ≥24 months and <18 years at screening
* Assent from patient and informed consent from parents/legal guardian

Exclusion Criteria:

* Uncertain diagnosis or variants of Alport syndrome such as a heterozygous carrier
* Alport syndrome levels III, or IV (albuminuria >300 mg/g Crea, creatinine clearance <60 mL/min, or end stage renal failure [ESRF])
* Known allergies or intolerances to ramipril or related compounds
* Known contraindication for ACEi-therapy
* Additional chronic renal, pulmonary or cardiac diseases
* Pregnancy and lactation

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2012-03; Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Time to next disease level | within 3 years
  Time to progression of Alport Syndrome to the next disease level within 3 years under ramipril treatment compared to placebo, for all randomised patients.
Incidence of Adverse Drug Events before progression | within 3 years
  Incidence of adverse drug events (ADEs, e.g., angioedema, acute renal failure, hyperkalaemia) under ramipril treatment before disease progression compared to placebo before disease progression, for all randomised patients.

SECONDARY OUTCOMES:
Albuminuria after three years | after 3 years
  Albuminuria after 3 years corrected for baseline albuminuria for patients randomised to receive ramipril compared to placebo.
Adverse Drug Events over three years | after 3 years
  Incidence of ADEs (e.g., angioedema, acute renal failure, hyperkalaemia) during 3 years of treatment for patients randomised to receive ramipril compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Gross, Prof., Study Chair — University Medical Center Goettingen, Department Nephrology and Rheumatology
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

REFERENCES:
- [Result] Gross O, Tonshoff B, Weber LT, Pape L, Latta K, Fehrenbach H, Lange-Sperandio B, Zappel H, Hoyer P, Staude H, Konig S, John U, Gellermann J, Hoppe B, Galiano M, Hoecker B, Ehren R, Lerch C, Kashtan CE, Harden M, Boeckhaus J, Friede T; German Pediatric Nephrology (GPN) Study Group and EARLY PRO-TECT Alport Investigators. A multicenter, randomized, placebo-controlled, double-blind phase 3 trial with open-arm comparison indicates safety and efficacy of nephroprotective therapy with ramipril in children with Alport's syndrome. Kidney Int. 2020 Jun;97(6):1275-1286. doi: 10.1016/j.kint.2019.12.015. Epub 2020 Jan 17. PMID 32299679
- [Derived] Kashtan CE, Gross O. Clinical practice recommendations for the diagnosis and management of Alport syndrome in children, adolescents, and young adults-an update for 2020. Pediatr Nephrol. 2021 Mar;36(3):711-719. doi: 10.1007/s00467-020-04819-6. Epub 2020 Nov 6. PMID 33159213
- [Derived] Boeckhaus J, Hoefele J, Riedhammer KM, Tonshoff B, Ehren R, Pape L, Latta K, Fehrenbach H, Lange-Sperandio B, Kettwig M, Hoyer P, Staude H, Konrad M, John U, Gellermann J, Hoppe B, Galiano M, Gessner M, Pohl M, Bergmann C, Friede T, Gross O; GPN Study Group and EARLY PRO-TECT Alport Investigators. Precise variant interpretation, phenotype ascertainment, and genotype-phenotype correlation of children in the EARLY PRO-TECT Alport trial. Clin Genet. 2021 Jan;99(1):143-156. doi: 10.1111/cge.13861. Epub 2020 Oct 25. PMID 33040356
- [Derived] Ahmed R, Duerr U, Gavenis K, Hilgers R, Gross O. Challenges for academic investigator-initiated pediatric trials for rare diseases. Clin Ther. 2014 Feb 1;36(2):184-90. doi: 10.1016/j.clinthera.2014.01.013. PMID 24529291
- See also: Related Information — http://www.alport.de